CLINICAL TRIAL: NCT06620263
Title: Ensuring Guideline Adherence and Cost Savings in Stress Ulcer Prophylaxis Practices in the Intensive Care Unit: a Pre-Post Education Study
Brief Title: Stress Ulcer Prophylaxis Practices in the Intensive Care Unit
Acronym: guideline
Status: Completed | Type: Observational
Sponsor: Yunus Emre AYHAN (Other)
Responsible Party: Sponsor-Investigator, Yunus Emre AYHAN, Specialist Clinical Pharmacist, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Organization: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Other Study IDs: 249/20.11.2023
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Stress Ulcer Prophylaxis
Keywords: Stress ulcer prophylaxis; Proton pump inhibitor; Intensive care unit; Clinical pharmacist

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pre-education period (PreEd): In PreEd, the SUP use of patients in the ICU was observed observationally for three months.
  Interventions: Other: Pre-education period (PreEd)
- Post-education period (PostEd): The SUP education program in the ICU was implemented for ICU physicians after examining the patient data in the first three months of the study. In the 3-month PostEd after the education program (April 3, 2024 - July 3, 2024), SUP was only used in patients in the ICU, and no intervention was observed. Throughout the study period, the appropriateness of SUP uses for the indication was evaluated according to the Sociedade Portuguesa de Cuidados (SPC) SUP guideline
  Interventions: Other: Post-education period (PostEd)

INTERVENTIONS:
Other: Pre-education period (PreEd) — No intervention. ). In PreEd, the SUP use of patients in the ICU was observed observationally for three months (January 1, 2024 - April 1, 2024).
  Groups: Pre-education period (PreEd)
Other: Post-education period (PostEd) — In the study, the SUP education program in the ICU was implemented for ICU physicians after examining the patient data in the first three months of the study. In the 3-month PostEd after the education program (April 3, 2024 - July 3, 2024), SUP was only used in patients in the ICU, and no intervention was observed.
  Groups: Post-education period (PostEd)

SUMMARY:
The present study aimed to examine the adherence of proton pump inhibitors (PPIs), commonly recommended for stress ulcer prevention (SUP) in patients in the intensive care unit (ICU), according to an international guideline. The objective of the study was to enhance the adherence of SUP prescriptions to the guideline, therefore preventing potential adverse effects and avoidable financial burden, and, consequently, attaining cost reduction.

DETAILED DESCRIPTION:
Background Intensive care unit (ICU) patients are prone to developing stress-related gastrointestinal (GI) bleeding, which is associated with increased morbidity and mortality. Respiratory failure, hypotension, coagulopathy, and especially prolonged mechanical ventilation (MV) are the most critical clinically significant risk factors for GI bleeding in patients. Many studies have shown that invasive MV for 48 hours or longer and coagulopathy are two independent risk factors for clinically significant upper GI bleeding in ICU patients.

Stress ulcer prophylaxis (SUP) is widely practiced in ICUs worldwide and is often (up to 70%) used inappropriately. Proton pump inhibitors (PPI) are among the most commonly used medications in critically ill patients for SUP. However, the inappropriate and quite inconsistent use of PPIs in ICUs has added unnecessary costs, enhanced risks related to adverse drug reactions, and possible complications like pneumonia, Clostridium difficile infections, hypomagnesemia, and bone fractures.

A few studies have assessed adherence with SUP guidelines and institutional standards under the surveillance of a pharmacist. The results of these studies implied that pharmacist supervision reduced the inappropriate use of SUP in patients and its associated healthcare costs. One of these studies noted that the intervention and adjustment of pharmacists reduced the incidence of inappropriate use of SUP and its associated costs from $26.75 and $2433 per 100 patient days pre-intervention to $7.14 and $239.80 per 100 patient days post-intervention with p<0.001. The same study emphasized that a comprehensive multidisciplinary approach must be implemented to decrease inappropriate SUP use in the ICU.

The aim of this study is to enhance adherence to the guidelines through an educational program focused on reducing inappropriate use of SUP in the ICU. The goal is to promote appropriate use of SUP based on indications, leading to cost savings.

Methods Study Design and Participants This study was designed as a non-randomized, controlled, prospective study created according to the pre-post education evaluation model. It was conducted in the anesthesia and reanimation ICU of a training and research hospital between January 2024 and July 2024 (6 months). The study was conducted in pre-education (PreEd) and post-education (PostEd). In PreEd, the SUP use of patients in the ICU was observed observationally for three months (January 1, 2024 - April 1, 2024). In the study, the SUP education program in the ICU was implemented for ICU physicians after examining the patient data in the first three months of the study. In the 3-month PostEd after the education program (April 3, 2024 - July 3, 2024), SUP was only used in patients in the ICU, and no intervention was observed. Throughout the study period, the appropriateness of SUP uses for the indication was evaluated according to the Sociedade Portuguesa de Cuidados (SPC) SUP guideline].

Education Program The education program was organized on April 3, 2024, after completing the 3-month PreEd review. The 1-hour education program was presented face-to-face to ICU physicians by a clinical pharmacist and an intensive care specialist physician. The content of the education included education on SUP, pathophysiology of stress ulcer, SUP risk/benefit situations, guidelines for SUP, introduction of appropriate SUP criteria according to the SPC SUP guideline, and frequently inappropriate SUP prescription situations in ICU, and the correct time to stop SUP. The evaluations obtained during the PreEd review in the ICU were also presented to the physicians participating in the education.

Data Collection Sociodemographic information, disease and medication history, existing laboratory values (coagulation parameters, procalcitonin, c-reactive protein, etc.), culture results, MV status, nutritional status, GI system bleeding status, pneumonia status, presence of Clostiridioides difficile, appropriate/inappropriate SUP use days and costs were obtained from the patient's treatment file and the hospital information management system with the utmost respect for personal privacy conditions.

Assessment of the Stress Ulcer Prophylaxis Use SUP use of ICU patients was evaluated throughout the week. SUP practices of ICU patients and patient data were reviewed by a clinical pharmacist and an intensive care specialist and evaluated for compliance with the SPC SUP criteria in terms of indication [12]. No intervention was made in the patients' SUP practices in either period.

Sample Size For the study's sample size, it was determined that there should be at least 42 patients in each period, based on the literature data that inappropriate SUP use in patient groups is reduced by approximately 30%, based on the calculation made on alpha 0.05 and 95% power values. Considering the 15% loss margin, it was decided to include 96 patients in the study, with at least 48 patients each period.

Definitions Authors defined significant GI bleeding as bleeding requiring a gastroscopy or blood transfusion upon clinician judgment. C. difficile infection was defined as the presence of relevant symptoms with positive fecal toxin and/or polymerase chain reaction in ICU patients after initiation of SUP in the ICU.

The rate of SUP use in appropriate indications was accepted as the percentage of PPIs used by a patient according to the SPC SUP guideline for the total number of hospital days.

Outcomes Measurement Adherence rates to SPC SUP guideline and costs of nonadherence were primary outcome measurements.

Inclusion and Exclusion Criteria Patients aged ≥18 years, those with an ICU stay longer than 24 hours, and those using PPIs for SUP were included in the study. Patients with a diagnosis of gastric cancer, history of GI, those with subtotal/total gastrectomy, those using PPIs for treatment indications such as dual antiplatelet therapy, and those admitted to the ICU with GI bleeding were excluded from the study.

Statistical analysis The study used descriptive statistics including mean, median, standard deviation, interquartile range (IQR), count, and percentages to show continuous variables' central tendency and variability. For categorical variables, frequency, and percentages were given. The Kolmogorov-Smirnov test was used to see if continuous variables followed the normal distribution. The result was non-parametric. The Mann-Whitney U tests were used to compare continuous variables between two groups. Categorical data was compared using Chi-square tests. A 95% confidence interval (CI) with a p-value less than 0.05 was considered statistically significant. Analysis of the dataset was done on an overall basis with the help of IBM SPSS Statistics for Windows, Version 29.0 (Armonk, New York: IBM Corp.), Cost Savings Analysis This study compared the costs of SUP agents prescribed for inappropriate indications between PreEd and PostEd. Finally, the SUP cost per patient was determined by multiplying the number of appropriate and inappropriate days of use in both PreEd and PostEd by the cost of PPI. Differences in the SUP costs between PreEd and PostEd are called cost-saving.

The costs for the SUP agents were estimated using current drug prices available from the hospital where this study was conducted. Thus, ten pantoprazole intravenous (IV) ampules were accepted for $3. Only the costs related to PPIs have been calculated. The calculation excluded nursing services and medical supplies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years,
* ICU stay longer than 24 hours,
* PPI use for SUP

Exclusion Criteria:

* Patients with a diagnosis of gastric cancer
* Patients with a history of gastrointestinal issues
* Individuals who have undergone subtotal or total gastrectomy
* Those using proton pump inhibitors (PPIs) for treatment indications such as dual antiplatelet therapy
* Patients admitted to the intensive care unit (ICU) with gastrointestinal bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This population includes ICU patients using PPI for SUP.
Sampling Method: Probability Sample
Enrollment: 495 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Stress ulcer prophylaxis appropriate rate | through study completion, an average of 1 year
  The appropriateness rates of SUP uses for the indication was evaluated according to the Sociedade Portuguesa de Cuidados (SPC) SUP guideline. Accordingly, the adherence rate was calculated by dividing the SUP prescriptions in accordance with the guideline during a patient's hospitalization by the SUP use during the entire hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu Şehir Hastanesi, Istanbul, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not have a legal right to share IPD in the country I am in. Therefore, I cannot share IPD.

REFERENCES:
- [Background] Mendes JJ, Silva MJ, Miguel LS, Goncalves MA, Oliveira MJ, Oliveira CDL, Gouveia J. Sociedade Portuguesa de Cuidados Intensivos guidelines for stress ulcer prophylaxis in the intensive care unit. Rev Bras Ter Intensiva. 2019;31(1):5-14. doi: 10.5935/0103-507X.20190002. Epub 2019 Feb 28. PMID 30843949
- See also: In this study, the guideline is the reference taken as the source for adherence. — https://pubmed.ncbi.nlm.nih.gov/30843949/